CLINICAL TRIAL: NCT06331832
Title: Treatment Guidelines for Expanded Access of Imvotamab (IGM-2323) in Patients With Relapsed/Refractory Non-Hodgkin Lymphomas From IGM-2323-001
Brief Title: Expanded Access of Imvotamab (IGM-2323) in Patients With R/R NHL
Status: No longer available | Type: Expanded Access
Sponsor: IGM Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2323-EAP; 2021-002339-44 (EudraCT Number)
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Relapsed/Refractory Non-Hodgkin Lymphomas
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: IGM2323 — Imvotamab is a recombinant monoclonal antibody of the IgM kappa isotype that targets the human CD20 antigen. Its component J-chain is fused to a single chain Fv antibody fragment which targets human CD3ε.

SUMMARY:
Expanded Access of Imvotamab (IGM-2323) in Patients with Relapsed/Refractory Non-Hodgkin Lymphomas from IGM-2323-001 clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrated clinical benefit (SD, PR, or CR) on clinical trial protocol IGM-2323-001
* There is no adequate alternative treatment available for the patient.
* Provided consent to continue treatment on expanded access program.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to the first dose.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use highly effective contraceptive measures.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use highly effective contraceptive.

Exclusion Criteria:

* History of severe allergic or anaphylactic reactions to mAb (or recombinant antibody related fusion proteins).
* Any medical condition or clinical laboratory abnormality likely to interfere with assessment of safety or efficacy of investigational product, or indicating patient would unlikely have potential benefit.
* Pregnant, breastfeeding, or intending to become pregnant during the program or within 2 months after the final dose of imvotamab.
* In the treating physician's judgement, the patient is unlikely to complete all procedures, including follow-up visits, or comply with the requirements for participation.
* Vaccination with live virus vaccines during treatment and for 3 months following the last cycle of Imvotamab.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (3):
- Sir Charles Gairdner Hospital, Nedlands, Western Australia, Australia
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea
- START-Madrid Centro Integral Oncologico Clara Campal, Madrid, Spain